CLINICAL TRIAL: NCT01238224
Title: The Effect of Selective PDE-5 Inhibition on Capillary Recruitment, Glucose Uptake and Endothelial Function Following a Mixed Meal in Patients With Type 2 Diabetes Patients.
Brief Title: Effects of PDE-5 Inhibition on Postprandial Hyperglycemia in Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Durability of study medications could not be guaranteed after the expire date.
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-003921-25
Record Dates: First submitted 2010-10-06; First posted 2010-11-10 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
Keywords: Insulin resistance; Phosphodiesterase-5 inhibition; Microdialysis; Type 2 diabetes; Endothelial dysfunction; Oral hypoglycaemic agents
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A single dose of placebo is administered 30 min before a mixed meal.
  Interventions: Drug: Tadalafil
- Tadalafil (Active Comparator): A single dose of tadalafil 20 mg is administered 30 min before a mixed meal.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — This is an acute study. Tadalafil 20 mg administered prior to a meal
  Other Names: Cialis

SUMMARY:
An increase of blood flow and capillary permeability decrease the impact of an endothelial barrier for glucose and insulin allowing them to reach their target cells in peripheral insulin sensitive organ in the human body. It is well known that insulin-resistant type 2 diabetes patients have an impaired blood flow in skeletal muscle and it is therefore important to elucidate means to reverse this metabolic defect.

The investigators have in a recently published study in type 2 diabetes patients used a drug against erectile dysfunction, the PDE-5 inhibitor tadalafil, with known effects on several vascular territories, to increase muscle blood flow in type 2 diabetes patients who were studied after fasting overnight.

The aim of this study is to test the hypothesis that tadalafil, compared to placebo, increases muscle glucose uptake and lowers blood glucose following a mixed meal served to type 2 diabetes patients.

DETAILED DESCRIPTION:
An increase of blood flow and capillary permeability decrease the impact of an endothelial barrier for glucose and insulin allowing them to reach their target cells in peripheral insulin sensitive organ in the human body. It is well known that insulin-resistant type 2 diabetes patients have an impaired blood flow in skeletal muscle and it is therefore important to elucidate means to reverse this metabolic defect.

The investigators have in a recently published study in type 2 diabetes patients used a drug against erectile dysfunction, the PDE-5 inhibitor tadalafil, with known effects on several vascular territories, to increase muscle blood flow in type 2 diabetes patients who were studied after fasting overnight. In fact, the investigators observed that tadalafil compared to placebo increased glucose uptake in muscle in parallel with an augmented capillary recruitment in muscle. This was the first publication to show that the pharmacological principle to inhibit the enzyme phosphodiesterase-5 (PDE-5) may mediate an increased muscle glucose uptake and, hence, may be a novel strategy to lower blood glucose in type 2 diabetes patients.

The aim of this study is to test the hypothesis that tadalafil, compared to placebo, increases muscle glucose uptake and lowers blood glucose following a mixed meal served to type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal state, defines as natural amenorrhea for at least 12 months.
2. Age; females 52-65 years, males: 40-65 years.
3. Type 2 diabetes based on fasting plasma glucose or 2-hr glucose after an OGTT.
4. Diabetes duration less than 5 years.

Exclusion Criteria:

1. Patients with concurrent use of nitrates or NO donors, history of heart or cerebrovascular disease, cardiac failure (stages NYHA II-IV), uncontrolled hypertension (> 160/100 mm Hg), significant diabetic complications, and inadequate glycemic control (HbA1c > 7%, ref value 3.5-5.3%)
2. Patients on glitazones, insulin, beta-blockers, ACE-inhibitors and corticosteroids

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Capillary recruitment, muscle glucose uptake and circulating glucose levels following a meal | Five hours after a mixed meal
  Capillary recruitment and glucose uptake in forearm muscle as well as circulating glucose levels following acute administration of tadalafil or placebo in type 2 diabetes patients.

SECONDARY OUTCOMES:
Vascular function and circulating biomarkers. | Five hours after a mixed meal
  Arterial stiffness as measured by pulse wave velocity and circulating concentrations of metabolic variables

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, MD, PhD, Principal Investigator — Region of Västra Götaland, Sahlgrenska University Hospital/Sahlgrenska University at University of Göteborg, Dept of Molecular and Clinical Medicine, SE 413 45 Göteborg, Sweden
Locations (1):
- The Wallenberg Laboratory, Dept of Molecular and Clinical Medicine, Sahlgrenska University Hospital, Bruna stråket 16,, Gothenburg, Sweden

REFERENCES:
- [Background] Jansson PA, Murdolo G, Sjogren L, Nystrom B, Sjostrand M, Strindberg L, Lonnroth P. Tadalafil increases muscle capillary recruitment and forearm glucose uptake in women with type 2 diabetes. Diabetologia. 2010 Oct;53(10):2205-8. doi: 10.1007/s00125-010-1819-4. Epub 2010 Jun 10. PMID 20535445